CLINICAL TRIAL: NCT02611011
Title: Assessing the Usability and Clinical Utility of the Congo Red Dot Test: A Survey
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 4005B
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Preeclampsia
Keywords: Congo Red Dot Test
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — urine samples collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women: Women seeking health services will perform the Congo Red Dot test (GV-005) individually by following the the test instructions
  Interventions: Device: Congo Red Test (GV-005)

INTERVENTIONS:
Device: Congo Red Test (GV-005) — The GV-005 is a simple test has been developed to detect unfolded or misfolded proteins in urine.

SUMMARY:
To determine if women can understand the instructions, carry out the test, and interpret the test results. Women will be recruited to complete a test instruction and comprehension assessment and a usability assessment.

DETAILED DESCRIPTION:
To determine if women can understand the instructions, carry out the test, and interpret the test results. Women will be recruited to complete a test instruction and comprehension assessment and a usability assessment. Study participants will be a convenience sample of women seeking health services. Participants will first be asked to review the instructions for the Congo Red Dot Test and complete a short written questionnaire that assesses their comprehension of the test instructions. Participants will then be asked to perform the test using a test control and to interpret the results obtained by answering a second written questionnaire. After the woman performs the test, a healthcare provider will use a matched control to perform a second test.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to consent for research
* Able to read Spanish well enough to read the test instructions
* Able to give informed consent

Exclusion Criteria:

* None

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women attending Centre de Salud Beatriz Velasco de Aleman for health services
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
CRD Test Comprehension | within 5 minutes of reading test instructions
  proportion of women who demonstrated various levels of understanding of the instructions for the CRD Test

SECONDARY OUTCOMES:
CRD Test Usability | within 5 minutes of performing test
  the proportion of women able to correctly use the CRD test

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, Dr, Principal Investigator — Gynuity Health Projects
Locations (1):
- Centro de Slaud Beatriz Velasco de Aleman, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided